CLINICAL TRIAL: NCT06986759
Title: Comparative Effects of Laser and Extracorpeal Shock Wave Therapy on Pain, Range of Motion and Function in Patients With Achilles Tendinopathy.
Brief Title: Comparative Effects of Laser and Extracorpeal Shock Wave in Patients With Achilles Tendinopathy.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0173
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-07-07 (Actual); Status verified 2025-07

CONDITIONS: Achilles Tendinopathy
Keywords: Pain; Function; Range of Motion
MeSH Terms: conditions — Pain | interventions — Lasers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser therapy protocol. (Active Comparator): The therapy system will be used the Thor DD Laser Therapy Unit. This will be a class 3B laser with an 810-nm, 100-mW infrared probe. Laser or placebo laser treatment protocols will be identical and will be delivered with the patients lying prone, with their foot over the end of the treatment plinth and the ankle plantar-grade. The contact method will be used to apply the laser treatment probe to 3 standardized points on both sides of the Achilles' tendon (6 in all: at the site of the lesion, 2cm proximal, and 2cm distal) for 30 seconds, giving a dose of 3J per point and 18J per session for the active probe. .
  Interventions: Other: Laser
- Extracorporeal shock wave therapy protocol. (Active Comparator): When treating Achilles tendinopathy, most researchers will be used 3 sessions of extracorporeal shock wave therapy (ESWT) with a one-week break in between. There will also be shorter breaks of 3 to 4 days or longer 2-week breaks. The number of pulses per session will range from 800 to 3000, and the pulse frequency will be between 4 and 50 Hz.
  Interventions: Other: Extracorporeal shock wave therapy protocol

INTERVENTIONS:
Other: Laser — The therapy system will be used the Thor DD Laser Therapy Unit. This will be a class 3B laser with an 810-nm, 100-mW infrared probe. Laser or placebo laser treatment protocols will be identical and will be delivered with the patients lying prone, with their foot over the end of the treatment plinth and the ankle plantar-grade. The contact method will be used to apply the laser treatment probe to 3 standardized points on both sides of the Achilles' tendon (6 in all: at the site of the lesion, 2cm proximal, and 2cm distal) for 30 seconds, giving a dose of 3J per point and 18J per session for the active probe(23). The treating physiotherapist, without any knowledge of which position on the switch will be the active laser, will select position 1 or 2 on the switch according to group allocation.
  Arms: Laser therapy protocol.
Other: Extracorporeal shock wave therapy protocol — When treating Achilles tendinopathy, most researchers will be used 3 sessions of extracorporeal shock wave therapy (ESWT) with a one-week break in between. There will also be shorter breaks of 3 to 4 days or longer 2-week breaks. The number of pulses per session will range from 800 to 3000, and the pulse frequency will be between 4 and 50 Hz.
  Arms: Extracorporeal shock wave therapy protocol.

SUMMARY:
Achilles tendinopathy is a prevalent condition characterized by pain, swelling, and impaired function of the Achilles tendon, commonly affecting athletes and active individuals. The disorder arises from a failed healing response, leading to degenerative changes in the tendon without significant inflammation. It is categorized into insertional (at the calcaneus-Achilles junction) and non-insertional (2-6 cm proximal to the insertion) types. Intrinsic risk factors include biomechanical abnormalities and systemic conditions like diabetes and hypertension, while extrinsic factors involve excessive mechanical load and training errors. Effective management of Achilles tendinopathy is crucial for preventing long-term disability and ensuring the continuation of physical activities.

DETAILED DESCRIPTION:
This study is a randomized clinical trial aimed at comparing the effectiveness of laser therapy and extracorporeal shock wave therapy on pain, range of motion, and function in patients with Achilles tendinopathy. The trial will be conducted at Hameed Latif Hospital, Lahore, Punjab, over a duration of nine months. A total of 44 participants, aged 18-40, diagnosed with Achilles tendinopathy and meeting specific inclusion criteria, will be randomly allocated into two groups using a lottery method. Group A will receive laser therapy, and Group B will undergo extracorporeal shock wave. Baseline and post-treatment measurements will be taken using the Visual Analogue Scale , Foot and Ankle Outcome Score , and goniometric measurements for range of motion. The data will be analyzed using SPSS software to evaluate the effectiveness of each treatment modality. For Group A, laser therapy will be administered using the Laser Therapy Unit, a class 3B laser with an 810-nm, 100-milliwatt infrared probe. The treatment will be applied to six standardized points around the Achilles tendon for 30 seconds each, providing a total dose of 18 joule per session. Group B will receive extracorporeal shock wave with each session involving 1500-3000 pulses at a frequency of 1-4 Hertz. Treatments will be conducted once a week for three weeks, with a one-week break between sessions. Both therapies aim to reduce pain and improve function by enhancing the healing processes of the damaged tendon.

ELIGIBILITY:
Inclusion Criteria:

* Age of patients 18-40.
* Diagnosed with chronic Achillis tendinopathy and NPRS rating more than 2.
* Both male and female.
* Patient must be diagnosed with Achillis Tendinopathy by single leg raise or Thompson test.

Exclusion Criteria:

* contraindications to LLLT to the area of the Achilles tendon.
* comorbid musculoskeletal or serious conditions that may have confounded treatment or anticipated recovery .
* nonsteroidal anti-inflammatory drug use steroid injections or surgery for the condition; insertional tendinopathy or bursitis (retrocalcaneal or Achilles; determined by clinical examination.
* neurologic signs; and adverse neural tension affecting the sciatic or sural nerve.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-07-24 (Estimated); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Numeric pain rating scale | 4 weeks
  The pain NPRS is a unidimensional measure of pain intensity, used to record patients' pain progression, or compare pain severity between patients with similar conditions. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. It has been shown that NPRS is valid, reliable and interval scale. NPRS has high test-retest reliability of ICC 0.98.

SECONDARY OUTCOMES:
Foot and ankle outcome | 4 weeks
  The FAOS is a patient-reported foot- and ankle-specific questionnaire including 42 items in 5 subscales evaluating pain, symptoms, function of daily living (ADL), function in sport and recreation (sport/rec), and quality of life (QOL). The outcome of FAOS is calculated based on a standardized scoring algorithm given a score between 0 and 100 for each of the 5 subscales. A score of 100 indicates the best possible results and 0 the worst outcome. Test-retest reliability shows intraclass correlation coefficient (95% confidence interval) was calculated as 0.94 (0.89-0.96

OTHER OUTCOMES:
Goniometer for range of motion | 4 weeks
  Goniometers are traditionally used to determine ROM of the ankle joint. Goniometers are considered valid and reliable clinical tools for assessing range of motion of joints of the extremities. A typical goniometric measurement of the ankle is made with the patient's leg supine on the treatment table and the fulcrum at the lateral malleolus whilst maintaining the bottom rod of the goniometer parallel with the tibia and fibula. the intraclass correlation coefficient (ICC) of ankle angle values were (dorsiflexion = 0.96), (plantarflexion = 0.81), (inversion = 0.92), (eversion = 0.95), (internal rotation = 0.92), and (external rotation = 0.78).

CONTACTS AND LOCATIONS:
Overall Officials: Muzna Munir, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Integrated Medical Care Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maffulli N, Longo UG, Kadakia A, Spiezia F. Achilles tendinopathy. Foot Ankle Surg. 2020 Apr;26(3):240-249. doi: 10.1016/j.fas.2019.03.009. Epub 2019 Apr 18. PMID 31031150
- [Background] Li HY, Hua YH. Achilles Tendinopathy: Current Concepts about the Basic Science and Clinical Treatments. Biomed Res Int. 2016;2016:6492597. doi: 10.1155/2016/6492597. Epub 2016 Nov 3. PMID 27885357
- [Background] Fares MY, Khachfe HH, Salhab HA, Zbib J, Fares Y, Fares J. Achilles tendinopathy: Exploring injury characteristics and current treatment modalities. Foot (Edinb). 2021 Mar;46:101715. doi: 10.1016/j.foot.2020.101715. Epub 2020 Jul 6. PMID 33039245
- [Background] von Rickenbach KJ, Borgstrom H, Tenforde A, Borg-Stein J, McInnis KC. Achilles Tendinopathy: Evaluation, Rehabilitation, and Prevention. Curr Sports Med Rep. 2021 Jun 1;20(6):327-334. doi: 10.1249/JSR.0000000000000855. PMID 34099611
- [Background] Wang Y, Zhou H, Nie Z, Cui S. Prevalence of Achilles tendinopathy in physical exercise: A systematic review and meta-analysis. Sports Med Health Sci. 2022 Mar 28;4(3):152-159. doi: 10.1016/j.smhs.2022.03.003. eCollection 2022 Sep. PMID 36090915
- [Background] Silbernagel KG, Hanlon S, Sprague A. Current Clinical Concepts: Conservative Management of Achilles Tendinopathy. J Athl Train. 2020 May;55(5):438-447. doi: 10.4085/1062-6050-356-19. Epub 2020 Apr 8. PMID 32267723
- [Background] Xergia SA, Tsarbou C, Liveris NI, Hadjithoma Mu, Tzanetakou IP. Risk factors for Achilles tendon rupture: an updated systematic review. Phys Sportsmed. 2023 Dec;51(6):506-516. doi: 10.1080/00913847.2022.2085505. Epub 2022 Jun 10. PMID 35670156
- [Background] van der Vlist AC, Winters M, Weir A, Ardern CL, Welton NJ, Caldwell DM, Verhaar JAN, de Vos RJ. Which treatment is most effective for patients with Achilles tendinopathy? A living systematic review with network meta-analysis of 29 randomised controlled trials. Br J Sports Med. 2021 Mar;55(5):249-256. doi: 10.1136/bjsports-2019-101872. Epub 2020 Jun 10. PMID 32522732
- [Background] Zhi X, Liu X, Han J, Xiang Y, Wu H, Wei S, Xu F. Nonoperative treatment of insertional Achilles tendinopathy: a systematic review. J Orthop Surg Res. 2021 Mar 30;16(1):233. doi: 10.1186/s13018-021-02370-0. PMID 33785026
- [Background] Brock-Jones K. The Effects of Low-Level Laser Therapy Versus Platelet Rich Plasma Therapy on Pain and Function in Patients with Achilles Tendinopathy: A Meta-Analysis: California State University, Fresno; 2023.